CLINICAL TRIAL: NCT06605677
Title: Knowledge Attitude and Practice Regarding Bloodstream Bacterial Infections and Antibiotics Usage Among Doctors in a Tertiary Hospital in Al Ain City, UAE: A Cross-Sectional Descriptive Study.
Brief Title: Knowledge Attitude and Practice Regarding Bloodstream Bacterial Infections and Antibiotics Usage Among Doctors.
Status: Enrolling by invitation | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Principal Investigator, Noura Saif Alnuaimi, Consutant Physician_ Internist, Abu Dhabi Health Services Company
Other Study IDs: HREC SEHA-IRB-559
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Bacteremia; Antimicrobial Stewardship; Antibiotic Use; Antibiotic Abuse
Keywords: bacteremia; antimicrobial resistance; antimicrobial stewardship; healthcare workers; antibiotic use; antibiotic abuse
MeSH Terms: conditions — Bacteremia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All doctors with valid medical license in Tawam and Al Ain Hospitals: The group excludes infectious disease physicians and microbiologists.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — An online questionnaire will be sent through e-mail to participants. It is divided into 4 sections: demography and general information 9 questions, knowledge 10 questions, attitude 10 questions and practice 10 questions. No previous similar studies were conducted in the United Arab Emirates (UAE) or internationally based on a search in PubMed and Cochrane library. Hence a validated questionnaire is lacking. Therefore, the questionnaire for this study is designed based on questions encountered daily by colleagues during the consultation, and it can serve the purpose of this study. Consent will be obtained and signed electronically by participants before starting the questionnaire. Participation involves minimal risk. Responses will be anonymous and confidential. Participants' involvement is voluntary, and they can withdraw at any time without any consequences. The time to complete the questionnaire is around 10-15 minutes. Each response will be saved using a unique identifier number.

SUMMARY:
This study is designed to use a questionnaire to assess doctors' knowledge, attitudes, and practices regarding bloodstream bacterial infections and antibiotic use in Tawam and Al Ain tertiary Hospitals (both hospitals have the same medical team) in Al Ain City, UAE.

DETAILED DESCRIPTION:
Background: Bloodstream bacterial infection is a serious medical problem and one of the leading causes of death worldwide among all age groups. Appropriate and early antibiotic use has been associated with better outcomes based on many clinical trials. On the other hand, misuse and abuse of antibiotics have been linked to long hospital stays, significant morbidity and mortality, increased medical costs and rising antimicrobial resistance (AMR). Statistics in hospitals involved in the study, showed increased antibiotic consumption compared to previous years and other regional healthcare facilities. Rates of AMR in the UAE have increased significantly in the last decade, based on the 2022 annual report.

Aims and objectives This study will assess knowledge, attitude and practice regarding bloodstream bacterial infections and antibiotics use among doctors. It is a questionnaire-based cross-sectional descriptive study that will be conducted at Tawam and Al Ain Hospitals (tertiary hospital, both hospitals have the same medical team).

The investigators want to explore the degree of knowledge and attitude, assess the appropriate usage of antibiotics among doctors in different subspecialties, assess any possible barriers, and find solutions such as medical education for this challenging medical problem.

ELIGIBILITY:
Inclusion Criteria:

All physicians with valid medical licenses working in Tawam and Al Ain tertiary hospitals

Exclusion Criteria:

Infectious diseases physicians and Microbiologists

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Licensed, practicing physicians, multinational
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Understanding physician knowledge on antibiotic use in bacterial bloodstream infections (bacteremia). | 1 year
  Questions to assess physicians' knowledge related to basic microbiology, bacterial infections and antibiotic spectrum of activity using dichotomous questions; yes/no.
Understanding physician attitude on antibiotic use in bacterial bloodstream infections (bacteremia). | 1 year
  Questions to assess physicians' attitude in bacteremia management using dichotomous questions; yes/no, Likert scale or multiple choices.
Understanding physician practices on antibiotic use in bacterial bloodstream infections (bacteremia). | 1 year
  Questions to assess physicians' practice in bacteremia management using dichotomous questions; yes/no, or multiple choices.

CONTACTS AND LOCATIONS:
Overall Officials: Noura Saif Alnuaimi, MD, Principal Investigator — Abu Dhabi Health Services Co-SEHA; Ahmed Al Hammadi, MD, Study Chair — Abu Dhabi Health Services Co-SEHA
Locations (1):
- Tawam and Al Ain Hospital, Al Ain City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomsen J et al. United Arab Emirates Surveillance of Antimicrobial Resistance Annual Report 2022.
- [Result] Labelle A, Juang P, Reichley R, Micek S, Hoffmann J, Hoban A, Hampton N, Kollef M. The determinants of hospital mortality among patients with septic shock receiving appropriate initial antibiotic treatment*. Crit Care Med. 2012 Jul;40(7):2016-21. doi: 10.1097/CCM.0b013e318250aa72. PMID 22584765
- [Result] Zahar JR, Timsit JF, Garrouste-Orgeas M, Francais A, Vesin A, Descorps-Declere A, Dubois Y, Souweine B, Haouache H, Goldgran-Toledano D, Allaouchiche B, Azoulay E, Adrie C. Outcomes in severe sepsis and patients with septic shock: pathogen species and infection sites are not associated with mortality. Crit Care Med. 2011 Aug;39(8):1886-95. doi: 10.1097/CCM.0b013e31821b827c. PMID 21516036
- [Result] Kreger BE, Craven DE, McCabe WR. Gram-negative bacteremia. IV. Re-evaluation of clinical features and treatment in 612 patients. Am J Med. 1980 Mar;68(3):344-55. doi: 10.1016/0002-9343(80)90102-3. PMID 6987871
- [Result] Bearman GM, Wenzel RP. Bacteremias: a leading cause of death. Arch Med Res. 2005 Nov-Dec;36(6):646-59. doi: 10.1016/j.arcmed.2005.02.005. PMID 16216646